CLINICAL TRIAL: NCT07321171
Title: Examining the Efficacy of a Stratified-Stepped-Care Model for Brief Interpersonal Couseling (IPC) in Youth With Imminent Suicidal Risk: A Prospective, Randomized Controlled Trial.
Brief Title: Stepped-Care for Suicidal Youth and Children
Acronym: SURE-CARE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shira Barzilay (Other)
Collaborators: Schneider Children's Medical Center, Israel (Other)
Responsible Party: Sponsor-Investigator, Shira Barzilay, Principal Investigator Dr Shira Barzilay, University of Haifa
Organization: University of Haifa (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0021-24-RMC; 2023/333 (Other Grant/Funding Number: The Israel national institute for health policy research)
Record Dates: First submitted 2025-09-28; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Suicidal Ideation and Behavior
Keywords: suicide prevention; youth; adolescent; inter personal counseling; stepped care; Suicide thoughts; paraprofessional; IPT; treatment
MeSH Terms: conditions — Suicidal Ideation; Behavior; Suicide Prevention | interventions — Interpersonal Psychotherapy

STUDY DESIGN:
Intervention Model Description: This study uses a parallel-group, randomized controlled trial (RCT) design. This means that after a baseline assessment, participants will be randomly assigned to one of two distinct, independent groups. Each group will receive a different intervention for the duration of the study, and their outcomes will be compared.
  The core of this model is the comparison between a novel, multi-layered treatment approach (Stratified Stepped-Care - SSC) and the existing standard of care (Care as Usual - CAU). The two groups are completely separate, with no participants switching between them. This design is robust for evaluating the effectiveness of a new intervention against an established one, as it minimizes bias and allows for a direct comparison of outcomes.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Although the therapists are aware of the type of treatment they are providing, the participants themselves are not aware of which research arm they belong to (the SSC group or the CAU group) at the time of allocation. They know that they are participating in a study to compare treatment methods, but the identity of the specific treatment they receive is only revealed to them upon the start of the treatment. This makes them "masked" for a certain period to prevent bias.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm: Stratified Stepped Care (SSC) (Experimental): The role of this arm is to test the efficacy of a new, tiered model for treating suicidal thoughts and behaviors (STB) in youth. Participants in this group will receive an intervention that is tailored to their specific needs and level of risk, as determined by an initial clinical assessment.
  Low-Intensity Treatment: Participants with mild-to-moderate STB will receive an adapted form of Interpersonal Counseling (IPC-A-SCI) delivered by a trained non-specialist. This intervention focuses on safety planning and improving interpersonal skills.
  High-Intensity Treatment: Participants with more severe STB, or those whose condition worsens, will receive Interpersonal Psychotherapy (IPT-A-SCI) from a professional therapist. This provides a clear "step-up" pathway to a more intensive level of care.
  Interventions: Behavioral: IPC-A-SCI (Interpersonal Counseling for Suicide Crisis Intervention); Behavioral: IPT-A-SCI (Interpersonal Psychotherapy for Adolescents with Suicidal Crisis Intervention)
- Control Arm: Care as Usual (CAU) (Active Comparator): The role of this arm is to serve as a comparison group to the SSC model. It represents the standard of care currently available in a public outpatient clinic in Israel.
  Standard Treatment: Participants in this arm will receive an initial psychiatric assessment. They will then be placed on a waitlist for a brief IPT intervention. Follow-up assessments will be conducted every three months. After completing the brief IPT, some participants may be referred to community services, and a small percentage may receive longer-term psychotherapy.
  Interventions: Behavioral: IPT-A-SCI (Interpersonal Psychotherapy for Adolescents with Suicidal Crisis Intervention)

INTERVENTIONS:
Behavioral: IPC-A-SCI (Interpersonal Counseling for Suicide Crisis Intervention) — The IPC-A-SCI is a manualized, low-intensity intervention adapted for adolescents experiencing suicidal thoughts and behaviors. It is based on Interpersonal Psychotherapy (IPT) principles but is designed to be delivered in a limited number of sessions by trained non-specialists. The protocol focuses on identifying and addressing interpersonal problems that may trigger or maintain suicidal behaviors. It includes core components such as safety planning, building interpersonal skills, and emotional processing, with a specific emphasis on involving parents in the treatment process. The intervention is a key component of the overall stratified stepped-care (SSC) model, which aims to provide targeted, effective, and accessible care in a public health setting.
  Arms: Intervention Arm: Stratified Stepped Care (SSC)
Behavioral: IPT-A-SCI (Interpersonal Psychotherapy for Adolescents with Suicidal Crisis Intervention) — The IPT-A-SCI is a crisis-focused psychotherapeutic intervention developed for adolescents with suicidal thoughts and behaviors. It is based on the principles of Interpersonal Psychotherapy (IPT).

SUMMARY:
The goal of this RCT study is to test the efficacy of a stratified stepped-care (SSC) model in reducing suicidal thoughts and behaviors (STB) in children and adolescents. The main questions it aims to answer are:

1. Does the SSC model effectively reduce STB and mental health symptoms?
2. Can the SSC model improve access to treatment and be cost-effective?

Researchers will compare the SSC model to Care as Usual (CAU). The SSC model includes low-intensity counseling delivered by non-specialists for mild STB and professional-delivered therapy for more severe cases. The CAU group will receive standard clinic treatment, which consists of a waitlist for brief therapy and follow-up.

Participants will be recruited from a clinic at Schneider Children's Medical Center, randomly assigned to either the SSC group or the CAU group, and Complete assessments at the start of the study and at 1, 3, and 6 months.

DETAILED DESCRIPTION:
Detailed Study Description This study is aimed at improving the care provided to children and adolescents experiencing suicidal thoughts and behaviors (STB). It addresses the significant public health challenge of rising suicide rates among youth and the systemic issues within mental health services, such as long waiting times and a shortage of professional staff. The research aims to develop a new, effective model of care that can be integrated into existing health systems.

The investigators will conduct a randomized controlled trial (RCT) comparing a new SSC model to the current standard of care, Care as Usual (CAU). The goal is to determine if the SSC model is more effective in reducing suicidal symptoms and improving mental health outcomes.

1. Provider Training:

   A key component of this model is the use of non-specialist mental health providers. The investigators will train a group of individuals, primarily psychology and community mental health graduate students with relevant experience, to deliver a low-intensity, evidence-based intervention. This intervention, Interpersonal Counseling for Suicidal Crisis Intervention (IPC-A-SCI), is a manualized protocol adapted for this study. The training will be conducted in a hybrid format (in-person and online), and the investigators will include weekly group supervision by a senior clinical psychologist. This training emphasizes the ethical and safety considerations necessary when working with this vulnerable population.
2. Participant Treatment and Data Collection:

Upon entering the study, senior clinicians will conduct a baseline assessment of each participant, including a diagnostic interview and a suicide risk evaluation. Participants will then be randomly assigned to one of two groups:

Intervention Group (SSC): Participants in this group will receive care based on their initial clinical assessment. Those with mild-to-moderate STB will receive the low-intensity IPC-A-SCI intervention from the newly trained non-specialist providers. If a patient's condition worsens, they can "step up" to a higher level of care, receiving brief IPT-A-SCI (Interpersonal Psychotherapy for Adolescents) from a professional therapist.

Control Group (CAU): Participants in this group will receive the standard treatment currently provided at the clinic. This typically involves an initial psychiatric assessment followed by placement on a waitlist for brief therapy.

Assessments to measure outcomes, including STB, depression, anxiety, and trauma, will be conducted at the beginning of the study and again at one, three, and six months. The investigators will analyze this data to compare the effectiveness of the two care models.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be between 6 and 18 years old, inclusive.
* Participants currently exhibit various forms of STB, including suicidal thoughts, gestures, behaviors, or attempted suicide.

Exclusion Criteria:

* Acute medical conditions.
* Current psychotic disorders.
* Non-fluency in Hebrew (language of intervention and assessment).
* Diagnosed intellectual disability.
* Diagnosed neurodevelopmental disorders (other than those that commonly co-occur with STB and are deemed manageable by the study team).
* Inability to provide informed consent (participant) or parental permission (parent/guardian).

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 350 (Estimated)
Dates: Start 2024-05-07 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Suicidal Thoughts and Behaviors (STB) as measured by the Columbia-Suicide Severity Rating Scale (C-SSRS). | Baseline, Week 4, Week 8, 12 Weeks Follow-up
  This primary outcome measure assesses the change in the severity of suicidal thoughts and behaviors (STB) among participants over time, relative to their initial state at baseline. Data for this measure will be collected using the Columbia-Suicide Severity Rating Scale (C-SSRS).
  The C-SSRS is a standardized, clinician-administered tool that consists of a series of questions designed to identify, classify, and quantify the severity of a person's suicidal thoughts and behaviors. The scale addresses five types of suicidal ideation (e.g., thoughts of suicide without a plan or intent) and six types of suicidal behaviors (e.g., actual suicide attempts).
  The assessment is conducted at multiple time points. The change in C-SSRS scores between these time points will be used to compare the intervention group with the control group, determining whether the new treatment is more effective in reducing suicidal risk in children and adolescents.
Feasibility of SSC Model Integration | From randomization up to one year after baseline.
  This measure evaluates the feasibility and fidelity of implementing the Stratified-Stepped-Care (SSC) model into the existing clinic workflow.
  Feasibility will be measured by calculating the percentage of adherence to the study protocol for both providers and participants (e.g., percentage of sessions completed, percentage of core protocol elements delivered). Fidelity will also be assessed via direct observation and completion of a standardized Protocol Adherence Checklist. Higher percentages indicate greater feasibility and fidelity to the SSC model and a better outcome.

SECONDARY OUTCOMES:
Depression: Measured by the Mood and Feelings Questionnaire (MFQ). | Baseline, Week 4, Week 8, 12 Weeks Follow-up
  This outcome measure assesses the change in depression levels among participants over time, relative to their initial state at baseline. Depression is measured using a standardized self-report questionnaire called the Mood and Feelings Questionnaire (MFQ).
  The MFQ is a standard tool for measuring the severity of depressive symptoms in children and adolescents. Participants are asked to rate the frequency of various depressive symptoms (such as feeling sad, hopeless, or losing interest in activities) on a rating scale. A higher score on the questionnaire indicates greater depression severity. The assessment is conducted at multiple time pointsץ
Total Cost of Mental Health Service Delivery per Participant | From randomization up to 6 months post-baseline.
  Costs in US Dollars will include direct service costs (e.g., provider salaries, training, supervision, facility costs) and indirect costs (e.g., costs associated with hospitalizations or emergency room visits related to STB). These components will be aggregated to provide a single value for the total cost of care for the study period.
  Lower total costs indicate greater economic efficiency and a better outcome.
Time (in Days) from Initial Intake to First Therapeutic Session | Initial Intake (Day 1) up up to first session of intervention
  The waiting time will be measured as the number of days from a participant's initial intake at the clinic to their first therapeutic session. This data will be collected for both the SSC group and the Care as Usual (CAU) group and will be compared to demonstrate whether the new model improves access.
  From Initial Intake (Day 1) through the start of the first therapeutic session for each participant.
  A lower number of days indicates reduced waiting time and a better outcome for access to care.
Change from Baseline in Anxiety Symptoms as measured by the Screen for Child Anxiety Related Emotional Disorders (SCARED). | Baseline, Week 4, Week 8, 12 Weeks Follow-up
  his outcome measure assesses the change in anxiety levels among participants over time, relative to their initial state at baseline. Anxiety is measured using a standardized self-report questionnaire called the Screen for Child Anxiety Related Emotional Disorders (SCARED).
  The SCARED is a standardized questionnaire that screens for five main types of anxiety disorders: panic disorder, generalized anxiety disorder, separation anxiety disorder, social anxiety, and school avoidance. Participants are asked to rate how true specific symptoms have been for them in the last three months, using a rating scale. A higher score on the questionnaire indicates greater anxiety severity.
Outcome Rating Scale (ORS) /Child Outcome Rating Scale (CORS) | Baseline, Week 4, Week 8, 12 Weeks Follow-up
  This measure assesses change across four domains: individual/personal functioning, interpersonal relationships, social role performance (e.g., school/work), and overall well-being.
  The Outcome Rating Scale (ORS) is for adolescents and their parents, and the Child Outcome Rating Scale (CORS) is for children ages 6-12 and their parents. Scores range from 0 to 40. (The scale consists of 4 items, scored from 0-10 each).
  Higher scores indicate better overall functioning, well-being, and progress in treatment.
Staff Survey of Acceptability (Adapted) | up to 1 year post initial training
  Satisfaction will be measured using a dedicated staff survey assessing the perceived ease of the training process, comfort level with the protocol, and perceived integration into clinic workflow.
  . Scores range from 1 to 5 (or the specific range of the Likert-type scale used).
  Higher scores indicate greater satisfaction with the training, supervision, and integration of the SSC model, reflecting a better outcome for implementation.
change in emotional and behavioral difficulties and prosocial strengths among participants. It is measured using the Strengths and Difficulties Questionnaire (SDQ), | Baseline, Week 4, Week 8, 12 Weeks Follow-up
  The questionnaire comprises five scales, each scored from 0 to 10: four difficulties scales (Emotional Symptoms, Conduct Problems, Hyperactivity/Inattention, and Peer Problems), and one Prosocial Strengths scale. The scores from the four difficulties scales are summed to create a Total Difficulties Score, ranging from 0 to 40. Higher scores on the four difficulties scales and the Total Difficulties Score indicate greater problems and a worse outcome. Conversely, higher scores on the Prosocial Strengths scale indicate greater positive behaviors and a better outcome.
the severity of Post-Traumatic Stress Disorder (PTSD) symptoms among participants. It is measured using the self-report questionnaire Child PTSD Symptom Scale (CPSS). | baseline
  This measure evaluates the change in the presence and severity of post-traumatic stress symptoms in participants using the Child Posttraumatic Stress Disorder Symptom Scale (CPSS). The CPSS is a reliable and well-known tool adapted for children and adolescents and is based on the DSM-5 diagnostic criteria for Post-Traumatic Stress Disorder (PTSD). Used to assess the presence and severity of symptoms consistent with the DSM-5 diagnostic clusters of PTSD.
  The questionnaire checks for the presence and severity of symptoms across four main clusters: Re-experiencing, Avoidance, Negative Alterations in Cognitions and Mood, and Hyperarousal. Scores range from 0 to 51. (27 items scored 0-4, with some items combined to yield a total score).
  Higher scores indicate greater severity of post-traumatic stress symptoms and a worse outcome.
Difficulties in Emotion Regulation Scale - State (DERS-State) | Baseline, Week 4, Week 8, 12 Weeks Follow-up
  This questionnaire assesses the current or recent experience of emotion regulation challenges across six key domains.
  Measures the presence and severity of emotion regulation difficulties in six Subscales Assessed 1. Non-acceptance of emotional responses: Rejects current emotional experiences.
  2. Difficulty engaging in goal-directed behavior: Difficulty concentrating or completing tasks when distressed.
  3. Lack of emotional awareness: Not paying attention to or understanding one's emotional state.
  4. Impulse control difficulties: Acting rashly or destructively when distressed.
  5. Lack of emotional clarity: Difficulty defining or distinguishing between different emotions.
  6. Limited access to emotion regulation strategies: Perceiving one's ability to cope as restricted.
  Scores typically range from 36 to 180 (based on the original 36-item full scale, with each item scored 1-5).
  Higher scores indicate greater difficulties in emotion regulation and a worse outcome.
The Deliberate Self-Harm Inventory (DASH-I), a self-report tool specifically designed for adolescents. | Baseline, Week 4, Week 8, 12 Weeks Follow-up
  This measure evaluates the frequency, types, and motives of Non-Suicidal Self-Injury (NSSI) using the Deliberate Attempt to Self-Harm Inventory (DASH-I). The DASH-I assesses various aspects of NSSI, including the types of behaviors (e.g., cutting, burning, hitting), their frequency, and the context and motives (e.g., to reduce emotional pain, punish oneself) behind the behaviors. Minimum Score: 0 (No NSSI episodes in the defined timeframe). Maximum Score: Varies, depending on the highest frequency category chosen (e.g., 50+).
  Higher scores on the frequency scales indicate more frequent self-harming behavior and a worse outcome.
  Since the DASH-I is an inventory, not a single psychometric scale, its maximum possible score is highly variable and often depends on the specific time frame assessed (e.g., past year).
The Children's Global Assessment Scale (CGAS) | Baseline, Week 4, Week 8, 12 Weeks Follow-up
  The Children's Global Assessment Scale (CGAS) used by the clinician to assess the participant's overall level of functioning and adaptation in daily life. Scores range from 1 to 100. Higher scores indicate better overall functioning. (100 = Superior functioning; 1 = Needs continuous supervision).
The Clinical Global Improvement (CGI) | Baseline, Week 4, Week 8, 12 Weeks Follow-up
  The Clinical Global Improvement (CGI) - Used by the clinician to assess the participant's severity of illness and improvement (or worsening) in symptoms over time. Scores range from 1 to 7. Lower scores indicate better/more significant improvement. (1 = Very much improved; 7 = Very much worse).
Client Satisfaction Questionnaire (CSQ-4) Score | immediately after the intervention
  This measure evaluates the acceptability and satisfaction of the SSC model from the perspective of the participants (children/adolescents and their parents). Scores range from 4 to 16 (4 items, scored 1-4 each).Higher scores indicate greater satisfaction with the intervention and a better outcome.
  Satisfaction levels of participants and their parents will be measured using the CSQ-4. The scores will be supplemented by qualitative data from brief verbal interviews (not scored as part of this specific outcome).

CONTACTS AND LOCATIONS:
Locations (1):
- Shneider children's Medical Center, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: Yes
The investigators plan to share de-identified Individual Participant Data (IPD) that underlie the results reported in this article, after de-identification. The data will be shared with researchers who provide a methodologically sound proposal and whose proposed use of the data has been approved by the study's scientific review committee or the institutional review board (IRB).
  Data will be available upon request to the Principal Investigator [Shira Barzilay, PhD], and will be delivered via a secured, password-protected electronic platform. Requestors will be required to sign a data access agreement (DAA) to ensure the protection of participant privacy and the sensitive nature of the data (suicide risk in minors). The data shared will include the research protocol, statistical analysis plan (SAP), and the anonymized dataset
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 6 months after the publication of the primary manuscript, for a period of 3 years following the initial release date.
Access Criteria: Access to the Individual Participant Data (IPD) will be granted only to qualified researchers outside of the immediate study team. Access requires that the requesting researcher submit a methodologically sound proposal for secondary analysis, and this proposal must be approved by the study's scientific review committee or the Institutional Review Board (IRB) to ensure the proposed use is ethical and aligned with participant consent. The following study documents and data will be made available:
  * De-identified Individual Participant Data (IPD)
  * Study Protocol
  * Statistical Analysis Plan (SAP)
  * Informed Consent Form (ICF) Access is contingent upon the requester signing a formal Data Access Agreement (DAA), which legally mandates adherence to privacy protocols and ensures protection of the sensitive nature of the data (suicide risk in minors).The de-identified dataset and supporting files will be delivered via a secured, password-protected electronic platform.